CLINICAL TRIAL: NCT03819244
Title: Clinical Comparison of The Use of Er,Cr:YSGG and Diode Lasers In Second Stage Implant Surgery
Brief Title: Comparison of Er,Cr:YSGG and Diode Lasers In Second Stage Implant Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Erkan Feslihan, Principal investigator, Yuzuncu Yil University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 24112017-01
Record Dates: First submitted 2019-01-16; First posted 2019-01-28 (Actual); Last update posted 2019-01-29 (Actual); Status verified 2019-01

CONDITIONS: Postoperative Pain; Soft Tissue Bleeding; Wound Heal
Keywords: Diode Laser; Erbium Laser; Second-stage Implant Surgery
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Diode laser (Experimental): Soft tissue incision with 940 nm Gallium Aluminum Arsenide diode laser, at implant recovery settings (2.5 W output power, average power: 1.25 W, pulse length : 1.00 ms, pulse interval: 1.00 ms) in second-stage implant surgery.
  Interventions: Device: 940 nm Gallium Aluminum Arsenide Diode Laser
- Erbium laser (Experimental): Soft tissue incision with 2780 nm Er,Cr:YSGG laser, at implant recovery settings (2.00 W power, 100 Hz, H mode, 10% water and 10% air) in second-stage implant surgery.
  Interventions: Device: 2780 nm Er,Cr:YSGG Laser

INTERVENTIONS:
Device: 940 nm Gallium Aluminum Arsenide Diode Laser — Exposure of the cover screw of osseointegrated dental implants embedded under oral mucosa by performing the soft tissue incision with diode laser for placing the healing abutment.
  Arms: Diode laser
Device: 2780 nm Er,Cr:YSGG Laser — Exposure of the cover screw of osseointegrated dental implants embedded under oral mucosa by performing the soft tissue incision with erbium laser for placing the healing abutment.
  Arms: Erbium laser

SUMMARY:
The study evaluates postoperative pain, intraoperative bleeding and wound healing after second stage implant surgery. Submerged implants were exposed with diode laser in Group 1 (n=20) and by using Er,Cr:YSGG laser in Group 2 (n=20).

ELIGIBILITY:
Inclusion Criteria:

* subject has osseointegrated implants embedded under oral mucosa.
* subject undergoes second-stage implant surgery.

Exclusion Criteria:

* inadequate keratinized gingiva in the implant site.
* localization of the implant site is not possible due to excessive thickness of the oral mucosa

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-11-27 (Actual); Primary Completion 2018-05-24 (Actual); Study Completion 2018-08-20 (Actual)

PRIMARY OUTCOMES:
Postoperative pain on 1st day | 1st Day
  Patients score pain intensity with numeric scale ranging between 0(no pain) to 10(most severe pain) on the postoperative 1st day. Pain scores on the postoperative 1st day in each group are compared.
Postoperative pain on 2nd day | 2nd Day
  Patients score pain intensity with numeric scale ranging between 0(no pain) to 10(most severe pain) on the postoperative 2nd day. Pain scores on the postoperative 2nd day in each group are compared.
Postoperative pain on 3rd day | 3rd Day
  Patients score pain intensity with numeric scale ranging between 0(no pain) to 10(most severe pain) on the postoperative 3rd day. Pain scores on the postoperative 3rd day in each group are compared.

SECONDARY OUTCOMES:
Number of analgesics used daily | 3 days
  Analgesic consumption per day on postoperative 1st, 2nd and 3rd days.
Intraoperative bleeding | During operation
  Bleeding during surgical procedure was scored by the physician as 1=minimal, 2=normal and 3=excessive bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Erkan Feslihan, DDS, Principal Investigator — Yuzuncu Yil University
Locations (1):
- Yuzuncu Yil University Faculty of Dentistry, Van, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be shared after publication of the article about this study.
Supporting Information: Study Protocol
Time Frame: Data will be available within 6 months.
Access Criteria: Open access

REFERENCES:
- [Background] El-Kholey KE. Efficacy and safety of a diode laser in second-stage implant surgery: a comparative study. Int J Oral Maxillofac Surg. 2014 May;43(5):633-8. doi: 10.1016/j.ijom.2013.10.003. Epub 2013 Nov 7. PMID 24210453
- [Background] Arnabat-Dominguez J, Espana-Tost AJ, Berini-Aytes L, Gay-Escoda C. Erbium:YAG laser application in the second phase of implant surgery: a pilot study in 20 patients. Int J Oral Maxillofac Implants. 2003 Jan-Feb;18(1):104-12. PMID 12608675

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-24): https://cdn.clinicaltrials.gov/large-docs/44/NCT03819244/Prot_SAP_000.pdf